CLINICAL TRIAL: NCT03330054
Title: Frequency Of Eye Problems In Type 2 Diabetes With Chronic Kidney Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mohammed Ramadan Abdallah (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Mohammed Ramadan Abdallah, Principal Investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: AssiutU MRAbdallah
Record Dates: First submitted 2017-10-31; First posted 2017-11-06 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Eye Diseases; Renal Impairment; Type2 Diabetes
MeSH Terms: conditions — Eye Diseases; Renal Insufficiency | interventions — Ophthalmoscopes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: 50 patients Type 2 Diabetes without renal impairment will be examined using fundoscope
  Interventions: Device: fundoscope
- Group B: 25 patients Type 2 Diabetes with chronic kidney disease not on replacement therapy (stage I-IV) will be examined using fundoscope
  Interventions: Device: fundoscope
- Group C: 25 patients Type 2 Diabetes with end stage renal disease on haemodialysis will be examined using fundoscope
  Interventions: Device: fundoscope

INTERVENTIONS:
Device: fundoscope — Fundoscope for eye examination

SUMMARY:
This study evaluate the frequency and type of eye problem among Type 2 Diabetics with renal impairment and effect of renal impairment and haemodialysis on diabetic retinopathy

DETAILED DESCRIPTION:
Chronic kidney disease is a descriptive term and is used for deteriorating kidney function of any underlying cause. Chronic kidney disease implies longstanding (>3 months), potentially progressive, impairment in renal function.(Kumar & Clark's ., 2016).

Diabetes mellitus is the most common cause of chronic kidney disease in developed countries. In patients with diabetes, there is a steady advance from microalbuminuria to dipstick positive proteinuria and a progression to renal failure. (Davidson's.,2014) .The most commonly diagnosed diabetes-related complications is diabetic retinopathy. Its prevalence increases with the duration of diabetes. Some 20%of people with type 1 diabetes will have retinal changes after 10 years, rising to >95% after20 years; 20-30% of people with type 2 diabetes have retinopathy at diagnosis.(Kumar & Clark's ., 2016) .

Also from risk factors of diabetic retinopathy is nephropathy, and if severe, is associated with worsening of Diabetic retinopathy. Conversely, treatment of renal disease (e.g. renal transplantation) may be associated with improvement of retinopathy and a better response to photocoagulation.(Kanaski ,2016) The high burden of ocular disease in Chronic kidney disease can be explained, in part, by the sharing of risk factors common to both kidney and eye diseases such as age, smoking, hypertension, diabetes, raised serum cholesterol and obesity. Ocular diseases may also be directly linked to chronic kidney disease via common pathogenic pathways, including, atherosclerosis, microangiopathy, inflammation and oxidative stress (Wong et al., 2014).

In our study we seek to do the following for participants :

1. A detailed history including

   1. Age, sex, smoking Habits
   2. Duration of diabetes mellitus and treatment.
   3. Chronic kidney disease stage by estimated glomerular filtration rate according to MDRD formula
   4. Duration of haemodialysis.
   5. Associated co-morbidity as hypertension,
   6. Therapeutic history eg; angiotensin converting enzyme, angiotensin II receptor blocker, amiodarone, erythropoietin.
2. Complete Clinical examination including haemodynamics, complete cardiac, chest, abdominal, lower limb examination, cranial nerve examination.
3. Complete eye examination including detailed fundus examination, classifying expected eye problems as:

   * Cataract. - Glaucoma
   * Cranial nerve affection
   * Retinopathy either proliferative, non proliferative or macular oedema.
4. The following investigations will be done:

   * Serum creatinine & Blood Urea for estimation of glomerular filtration rate
   * Glycated haemoglobin (HbA1c).
   * lipogram.
   * Complete blood count
   * ECG

ELIGIBILITY:
Inclusion Criteria:

* 50 patients Type 2 Diabetes without renal impairment.
* 25 patients Type 2 Diabetes with chronic kidney disease not on replacement therapy. (stage I-IV)
* 25 patients Type 2 Diabetes with end-stage renal disease on haemodialysis

Exclusion Criteria:

* patients with previous history of eye problems and any systemic disease.
* Type 1 Diabetics .
* Acute kidney injury in Diabetics.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Group A 50 patients Type 2 Diabetes without renal impairment. from outpatient clinic Group B 25 patients Type 2 Diabetes with chronic kidney disease not on replacement therapy. (stage I-IV) from outpatient clinic and admitted patient in Luxor International Hospital.
  Group C 25 patients Type 2 Diabetes with end-stage renal disease on haemodialysis from Haemodialysis unit in Luxor International Hospital.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-12-01 (Estimated); Primary Completion 2018-05-01 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
Frequency Of Eye problems In Type 2 Diabetes with Chronic Kidney Disease | 2 days for each participant to be assessed
  To evaluate the frequency and type of eye problem among:
  1. Type 2 Diabetics not having renal impairment.
  2. Type 2 Diabetics with chronic kidney disease not on replacement therapy.
  3. Type 2 Diabetics with end stage renal disease on haemodialysis.

CONTACTS AND LOCATIONS:
Overall Officials: Lobna F El-Toony, MD, Study Chair — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided